CLINICAL TRIAL: NCT01265004
Title: Evaluation of Microcirculation in Skin and Tendon After Surgical Treatment of Acute Rupture of the Achilles Tendon With Stitches or Fibrin-glue
Brief Title: Identification of Microcirculation After Surgical Treatment of Rupture of the Achilles Tendon
Acronym: MicroASR
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC-A10-26
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Microcirculation; Achilles Tendon Rupture
Keywords: Functional outcome
MeSH Terms: interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Stitches, rupture of achilles tendon: Patients, in who the achilles tendon rupture was treated with tendon surgery including a special way of stitching to preserve the sliding ability of the tendon.
  Interventions: Procedure: Stitches
- Fibrin-glue, rupture of achilles tendon: Patients, who received a surgical treatment including a fixing of the tendon with fibrin-glue.
  Interventions: Procedure: Fibrin-glue
- Stiches and Fibrin-glue: Patients, in who the achilles rupture was treated with stitches and fibrin-glue.
  Interventions: Procedure: Stitches and Fibrin-glue

INTERVENTIONS:
Procedure: Stitches — Surgical treatment of a rupture of the achilles tendon, in which both end are fastened with a U-forming stitching
  Groups: Stitches, rupture of achilles tendon
Procedure: Fibrin-glue — Surgical treatment, in which both ends are glued together using a medical fibrin-containing glue
  Groups: Fibrin-glue, rupture of achilles tendon
Procedure: Stitches and Fibrin-glue — Surgical treatment, in which both ends of the ruptured tendon are fastened together with u-forming stitches as well as fibrin-glue
  Groups: Stiches and Fibrin-glue

SUMMARY:
This project investigates microcirculation in skin and tendon after a rupture of the Achilles tendon. Three different treatments are compared: stitches of the tendon, fibrin-glue and the combination of both.

DETAILED DESCRIPTION:
This project investigates microcirculation in skin and tendon after a rupture of the Achilles tendon. Three different treatments are compared: stitches of the tendon, fibrin-glue and the combination of both.

Every method is long established and can be treated as clinical equal. So the surgical treatment is chosen randomly for each patient.

For this cause the microcirculation is registered by O2c, which works with measuring reflected lightwaves. It is strictly noninvasive and causes absolutely no pain for the patient. The measurement device consists of two small probes, which simply stick to the patient´s skin. There are nine measurements on this study: one before and one shortly after the surgery, followed by three measuring appointment every 6 hours (6,12,18,24 h post-op).Afterwards there are appointments planed after 12 days and 6 month. On the last appointment the patients are questioned according to established scores like AOFAS or VAS to register the functional outcome and level of pain.

Clinical parameters like time between rupture and surgical treatment, hospitalisation time, and form of anaesthesia are included to create comparable patient profiles. After 6 moths the last measurement appointment is stated, in which the clinical outcome is registered by Scores, e.g Mann-Whitney-Wilcoxon-Test.

This study is to detect any difference in wound heeling, re-rupture rate and functionality between these three methods.

ELIGIBILITY:
Inclusion Criteria:

* Acute rupture of the achilles tendon (on one or both sides)
* Older than 18 year of age
* Firmed letter of approval
* Patient speaks/understands German
* Planed surgical treatment
* No more than 48h after rupture

Exclusion Criteria:

* No-traumatic rupture of the achilles tendon
* More than 48h after rupture
* No planed surgical treatment
* History of surgery on the injured leg
* Condition of diabetes mellitus
* Condition of peripheral artery occlusive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute traumatic rupture of the achilles tendon
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Microcirculation | 6 month
  The microcirculation is measured by O2c, an non-invalive device functioning with lightwaves. Based on this data the soft tissue damage, edema and healing process is protocoled.

SECONDARY OUTCOMES:
Functional outcome | 6 month
  After 6 month the functinal outcome is measured by clinical scores.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Pape, Univ-prof.MD, Study Chair — Chief of medicine
Locations (1):
- Universal Hospital of the RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany